CLINICAL TRIAL: NCT01241786
Title: A Phase II, Single Arm Study Examining the Combination of Revlimid (Lenalidomide) and Vidaza (Azacitidine) (RA-CLL) for the Treatment of Relapsed/Refractory Chronic Lymphocytic Leukemia (CLL) and Small Lymphocytic Lymphoma (SLL)
Brief Title: Study Examining the Combination of Revlimid (Lenalidomide)and Vidaza (Azacitidine) for Relapsed/Refractory CLL and SLL
Acronym: VZCLLPI0146
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was closed early due to poor accrual
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00001361
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Results first posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-06

CONDITIONS: Chronic Lymphocytic Leukemia(CLL); Small Lymphocytic Lymphoma
Keywords: chronic lymphocytic leukemia (CLL); Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- response to Vidaza + Revlimid (Experimental): response to combination of azacitidine + lenalidomide A Phase II, Single Arm Study Examining the Combination of Revlimid (Lenalidomide) and Vidaza (Azacitidine) (RA-CLL) for the Treatment of Relapsed/Refractory Chronic Lymphocytic Leukemia (CLL) and Small Lymphocytic Lymphoma (SLL)
  Interventions: Drug: Revlimid; Drug: Azacitidine

INTERVENTIONS:
Drug: Revlimid — Lenalidomide PO daily Day 1-21. For patients with baseline calculated creatinine clearance ≥ 30 ml/min and < 60 ml/min the starting dose is 5 mg every other day (odd numbered days during Days 1-21). For patients with baseline calculated creatinine clearance ≥ 60 ml/min the starting dose is 5 mg daily on Days 1-21).
  Other Names: Lenalidomide
Drug: Azacitidine — Azacitidine 75 mg/m2 IV or SC D 1-5
  Other Names: Vidaza

SUMMARY:
To determine the response to the combination of Revlimid (Lenalidomide)+ Vidaza (Azacitidine) in patients with relapsed/refractory CLL and SLL

Hypothesis- lenalidomide's activity in combination with azacitidine may further enhance its activity and the durability of treatment response.

DETAILED DESCRIPTION:
Treatment response of lenalidomide's activity in combination with azacitidine may further enhance its activity and the durability of treatment response.

ELIGIBILITY:
Inclusion Criteria:

Patients must be age ≥ 18 must have an ECOG PS ≤ 2 must understand and voluntarily sign informed consent adhere to the study protocol requirements and schedule must carry the diagnosis of B-CLL/SLL, SLL/CLL must be defined as relapsed or refractory disease Pts. must have received and failed at least one purine-based treatment regimen (ie. FCR, FR, PCR, Fludarabine) or alemtuzumab-based regimen or bendamustine-based regimen prior to study enrollment Serum bilirubin levels <1.5 times the upper limit of the normal range for the laboratory (ULN) Higher levels are acceptable if these can be attributed to active hemolysis, ineffective erythropoiesis or Gilbert's disease.Serum (SGOT) [AST])(SGPT) [ALT]) levels <2 x ULN or <5 x ULN if hepatic metastases are present) Subjects must have calculated creatinine clearance ≥ 30ml/min Absolute neutrophil count > 1.0 x 109 / L Platelet count > 50x 109 / L (unless bone marrow is heavily infiltrated with underlying disease (50% or more) Disease free of prior malignancies for > 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast All participants must be registered into the mandatory RevAssist® program Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin) Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours prior to prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.

Exclusion Criteria: - Patient must not have any serious medical condition, laboratory abnormality, or psychiatric illness that would places the subject at unacceptable risk or confound the interpretation of data from the study Patients must be lenalidomide / azacitidine naïve prior to study enrollment Patients must not be HIV, Hepatitis B or Hepatitis C positive, except for Patients who are seropositive because of hepatitis B virus vaccine are eligible Patients must not have received chemotherapy, immunotherapy or any experimental study drug for CLL or SLL at least 4 weeks prior to study enrollment and initiation of treatment Patients with history of B-CLL and the development of prolymphocytic leukemia or Richter's transformation Known or suspected hypersensitivity to azacitidine, mannitol, thalidomide or Lenalidomide Pregnant or breast feeding females are not eligible or lactating females must agree not to breast feed while taking Lenalidomide Evidence of laboratory TLS by Cairo-Bishop Definition of Tumor Lysis Syndrome Subjects may be enrolled upon correction of electrolyte abnormalities Patients with advanced malignant hepatic tumors; Concurrent use of other anti-cancer agents or treatments, or Uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Mato, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of five subject participated in the trial.
Pre-assignment Details: A total of five patients were screened and consented for study and scheduled to start cycle 1
Groups:
- Revlimid (Lenalidomide)and Vidaza (Azacitidine): Study Examining the Combination of Revlimid (Lenalidomide)and Vidaza (Azacitidine) for Relapsed/Refractory CLL and SLL.
Period: Overall Study
Arm/Group | Revlimid (Lenalidomide)and Vidaza (Azacitidine)
Started | 5
Completed | 0
Not Completed | 5
Not completed — Lack of Efficacy | 5

BASELINE CHARACTERISTICS:
Population: A total of five subject participated in the trial. The study was closed early due to poor accrual on 8/17/2011 - the primary endpoint was not met, therefore there are no results to report as we do not have the power to answer the primary question.
Groups:
- Revlamid + Vidaza: The study was closed early due to poor accrual on 8/17/2011 - therefore we do not have the power to answer the primary question.
Arm/Group | Revlamid + Vidaza
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: the Rate of Response to the Combination of Azacitidine + Lenalidomide in Select Patients
Description: the rate of response to the combination of azacitidine + lenalidomide in select patients with relapsed/refractory CLL and small lymphocytic lymphoma (SLL).
Time Frame: 9 Months
Population: Zero patients achieved a response to the combination
Measure: Number; unit: participants
Groups:
- Study Terminated: Study terminated - closed early
Arm/Group | Study Terminated
Number analyzed (Participants) | 5
participants | 0

2. Secondary Outcome: Assess for Treatment Related Toxicity Following Administration of Lenalidomide/ Azacitidine.
Time Frame: 30 days after treatment completion (up to 10 Months)
Measure: Number; unit: participants
Arm/Group | Revlamid + Vidaza
Number analyzed (Participants) | 5
participants | 1

3. Secondary Outcome: The Progression Free Survival of Patients Treated With the Combination of Lenalidomide and Azacitidine
Time Frame: 9 Months
Measure: Median (Full Range); unit: Months
Arm/Group | Revlamid + Vidaza
Number analyzed (Participants) | 4
Months | 1 [1 to 2.5]

4. Secondary Outcome: The Overall Survival of Patients Treated With the Combination of Lenalidomide and Azacitidine
Time Frame: 9 Months
Measure: Number; unit: participants
Arm/Group | Revlamid + Vidaza
Number analyzed (Participants) | 5
participants | 5

ADVERSE EVENTS:
Groups:
- Revlimid + Vidaza: Drug: Revlimid Lenalidomide PO daily Day 1-21. For patients with baseline calculated creatinine clearance ≥ 30 ml/min and < 60 ml/min the starting dose is 5 mg every other day (odd numbered days during Days 1-21). For patients with baseline calculated creatinine clearance ≥ 60 ml/min the starting dose is 5 mg daily on Days 1-21).
  Other Names:
  Lenalidomide Drug: Azacitidine Azacitidine 75 mg/m2 IV or SC D 1-5
  Other Names:
  Vidaza
Arm/Group | Revlimid + Vidaza
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Revlimid + Vidaza (N=5)
Syncope (Nervous system disorders) | 1 (1)
Pelvic Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Disease Progression (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
Five patients were screened, consented and started cycle 1 but all patients were removed from study due to non response. The study was closed early due to poor accrual on 8/17/2011 before completing the timeframe required for statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes